CLINICAL TRIAL: NCT00297063
Title: Clinical Evaluation of Rosiglitazone Malate (BRL49653C) in Patients With Type 2 Diabetes Mellitus (Monotherapy) - Double-Blind Comparative Study of Rosiglitazone Maleate vs. Pioglitazone Hydrochloride and Placebo -
Brief Title: BRL49653C In Type 2 Diabetes -Comparison Study With Pioglitazone And Placebo By Monotherapy-
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: AVD104742
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: rosiglitazone; vandia; Type 2 diabetes mellitus; diabetes;
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
This study is designed to compare the efficacy and safety of BRL49653C versus pioglitazone and placebo.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes mellitus.
* Managed by diet therapy.
* Must have adequate blood, liver and kidney function.

Exclusion criteria:

* Serious cardiovascular disease or serious hepatic disease.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2006-01-11 (Actual); Primary Completion 2007-05-31 (Actual); Study Completion 2007-05-31 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline at Week 28. | 28 Weeks

SECONDARY OUTCOMES:
Efficacy variables (changes from baseline in FPG, fasting insulin, HOMA-IR and HOMA-beta) at stipulated date in each treatment group. | 28 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Japan (11):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kikuchi M, Kaku K, Odawara M, Momomura S, Ishii R. Efficacy and tolerability of rosiglitazone and pioglitazone in drug-naive Japanese patients with type 2 diabetes mellitus: a double-blind, 28 weeks' treatment, comparative study. Curr Med Res Opin. 2012 Jun;28(6):1007-16. doi: 10.1185/03007995.2012.694361. Epub 2012 Jun 6. PMID 22587483
- [Background] MacDonald MR, Petrie MC, Home PD, Komajda M, Jones NP, Beck-Nielsen H, Gomis R, Hanefeld M, Pocock SJ, Curtis PS, McMurray JJ. Incidence and prevalence of unrecognized myocardial infarction in people with diabetes: a substudy of the Rosiglitazone Evaluated for Cardiac Outcomes and Regulation of Glycemia in Diabetes (RECORD) study. Diabetes Care. 2011 Jun;34(6):1394-6. doi: 10.2337/dc10-2398. Epub 2011 May 11. PMID 21562320
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: AVD104742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVD104742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVD104742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVD104742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVD104742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVD104742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVD104742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register